Title: A Phase 2a, Multi-center, Double-blind, Placebo-controlled Study Evaluating ABI-H0731 + Entecavir vs Entecavir Alone for the Treatment of Viremic, HBeAg-positive Patients with Chronic Hepatitis B

NCT number: NCT03577171

Date: 6 August 2019

Statistical Analysis Plan Version Date; Final v1.0 06Aug2019

# Statistical Analysis Plan

| Sponsor: | Assembly Biosciences |
|---|---|
| Protocol No: | ABI-H0731-202 |
| PRA Project Id: | ASM31202-731202 |
| Protocol Version: | Amendment 1 v2.1 / 30 July 2018 (UK only) Amendment 1 v2.0 / 18 June 2018 (USA, Canada, NZ, HKG) Original v1.0 / 15 May 2018 |

| Title: | A Phase 2a, Multi-center, Double-blind, Placebo-controlled Study Evaluating ABI-<br>H0731+Entecavir vs Entecavir Alone for the Treatment of Viremic, HBeAg-positive<br>Patients with Chronic Hepatitis B |
|---|---|
| CRF Version Date: | 25 September 2018 |
| SAP No./Date | Final v1.0 / 06 Aug 2019 . |

## 1.0 Approvals

| Sponsor: Assembly Bios | sciences |
|----------------------------------|----------|
| Representative/ Title: | |
| Signature /Date: | |
| Representative/ Title: | |
| Signature /Date: | |
| PRA | |
| Project Manager/Title: | |
| Signature /Date: | |
| Biostatistician / Title (Owner): | |
| Signature /Date: | |

Statistical Analysis Plan Version Date: Final v1.0 06Aug2019

## **Statistical Analysis Plan**

| Sponsor: | Assembly Biosciences |
|---|---|
| Protocol No: | ABI-H0731-202 |
| PRA Project Id: | ASM31202-731202 |
| Protocol Version: | Amendment 1 v2.1 / 30 July 2018 (UK only) Amendment 1 v2.0 / 18 June 2018 (USA, Canada, NZ, HKG) Original v1.0 / 15 May 2018 |

| Title: | A Phase 2a, Multi-center, Double-blind, Placebo-controlled Study Evaluating ABI-H0731+Entecavir vs Entecavir Alone for the Treatment of Viremic, HBeAg-positive Patients with Chronic Hepatitis B |
|---|---|
| CRF Version Date: | 25 September 2018 |
| SAP No./Date | Final v1.0 / 06 Aug 2019 |

## 1.0 Approvals

| Sponsor: Assembly Bio | sciences | |
|-----------------------|----------|---|
| Signature /Date: | | |
| Signature /Date: | | |
| PRA | | |
| Signature /Date: | | • |
| Signature /Date: | | |

PRS 005 T 17 G 

## Statistical Analysis Plan

#### Version Date: Final v1.0 06Aug2019

## **Table of Contents**

| 1.0 Approvals | 1 |
|-----------------------------------------------------|----------|
| Table of Contents | 2 |
| 2.0 Purpose | 4 |
| 3.0 Scope | 4 |
| 4.0 Introduction | 4 |
| 4.1 Changes from Protocol | 4 |
| 5.0 Study Objectives | 4 |
| 5.1 Primary Objectives | 4 |
| 5.2 Secondary Objectives | 5 |
| 5.3 Exploratory Objectives | 5 |
| 6.0 Study Design | 5 |
| 6.1 Sample Size Considerations | <i>6</i> |
| 6.2 Randomization | 6 |
| 6.3 Schedule of Assessments | <i>6</i> |
| 7.0 Study Endpoints, Variables and Covariates | 10 |
| 7.1 Efficacy Endpoints and Variables | 10 |
| 7.1.1 Primary Efficacy Endpoints | 10 |
| 7.1.2 Secondary Endpoints | |
| 7.1.3 Exploratory Efficacy Endpoints | 10 |
| 7.2 Safety Endpoints and Variables | 11 |
| 7.2.1 Adverse Events | 11 |
| 7.2.2 Clinical Laboratory Tests | 12 |
| 7.2.3 Vital Signs | 13 |
| 7.2.4 12-Lead ECG | |
| 7.3 Pharmacokinetic Endpoints and Variables | 14 |
| 7.4 Other Variables | 14 |
| 7.5 Predetermined Covariates and Prognostic Factors | 15 |
| 8.0 Definitions | 15 |
| 9.0 Analysis Sets | 15 |
| 9.1 Intent-to-Treat | |
| 9.2 Safety | 15 |
| 9.3 Pharmacokinetic | |
| 9.4 Pharmacogenomic | 16 |
| 10.0 Interim Analyses | 16 |
| 10.1 Week 4 Pharmacokinetic Analysis | 16 |
| 10.2 Week 12 Safety Analysis | 17 |
| 11.0 Data Review | 17 |
| 11.1 Data Handling and Transfer | 17 |
| 11.2 Data Screening | |
| 12.0 Statistical Methods | |
| 12.1 General Considerations | |
| 12.2 Handling of Missing Data / Imputation Methods | 18 |
| 12.3 Subject Disposition | 20 |
| 12.4 Protocol Deviations | |
| 12.5 Demographic and Baseline Characteristics | |
| 12.6 Treatments | 21 |

#### Statistical Analysis Plan

Version Date: Final v1.0 06Aug2019

| 12.6.1 Prior and Concomitant Medications | 21 |
|---|---|
| 12.6.2 Procedures | 22 |
| 12.6.3 Compliance and Exposure to Study Drug | 22 |
| 12.7 Efficacy Analyses | 22 |
| 12.7.1 Primary Endpoint Assessment: HBV DNA Change from Baseline | |
| 12.7.2 Secondary and Exploratory Assessments | |
| 12.8 Safety Analyses | 25 |
| <b>12.8 Safety Analyses</b> 12.8.1 Adverse Events | 25 |
| 12.8.2 Deaths and Serious Adverse Events | 26 |
| 12.8.3 Central Laboratory Data | |
| 12.8.4 Vital Signs | |
| 12.8.5 Physical Examinations, ECGs, and Other Observations Related to Safety | |
| 12.9 Pharmacokinetics | |
| 13.0 Validation | 28 |
| 14.0 References | 28 |
| Appendix 1 Glossary of Abbreviations | 29 |
| Appendix 2 Tables, Figures, Listings, and Supportive SAS Output Appendices | |
| Appendix 3 Grading of Laboratory Values | |
| Laboratory Values*: Chemistries | |
| Hematology | 35 |
| Urinalysis | 36 |
| ~ <i>y</i> ~ | |



Statistical Analysis Plan


## 2.0 Purpose

The Statistical Analysis Plan (SAP) describes the statistical methods to be used during the reporting and analyses of data collected under Assembly Biosciences Protocol ABI-H0731-202, "A Phase 2a, Multicenter, Double-blind, Placebo-controlled Study Evaluating ABI-H0731 + Entecavir vs Entecavir Alone for the Treatment of Viremic, HBeAg-positive Patients with Chronic Hepatitis B".

## 3.0 **Scope**

This plan is a living document that will be created during the trial start-up. The Statistical Analysis Plan will be drafted within three months of final CRF and maintained throughout the lifecycle of the trial. Each version of the SAP will require sign off from the Project Manager and the Sponsor representatives prior to programming starting or being updated as a result of an amended version of the SAP.

The SAP outlines the following:

- Study objectives
- Study design
- Variables analyzed and analysis sets
- · Applicable study definitions
- Statistical methods regarding important protocol deviations, study drug exposure, efficacy analysis, concomitant medications, adverse events handling, laboratory data and physical examinations

#### 4.0 Introduction

This SAP should be read in conjunction with the study protocol and case report form (CRF). This version of the plan has been developed using the Protocol Amendment 1.0, v2.1 dated 30 July 2018 and CRF dated 30 August 2018. Any further changes to the protocol or CRF may necessitate updates to the SAP.

Versions of the SAP up to Sponsor approval will be known as a draft SAP. If necessary, changes following final approval of the SAP will be tracked in a SAP Change Log. The final sponsor approval of any amended version of the SAP will occur prior to database lock.

## 4.1 Changes from Protocol

Following an increase in the number of subjects in the sister protocol ABI-H0731-201 (Study 201), the timing of DMC meetings was changed to accommodate the two protocols in a single programmatic overview. As a result, instead of requiring all subjects in Study 202 (and separately in Study 201) to have completed Week 12 prior to triggering a DMC, the DMC trigger was 25% of subjects across BOTH studies completing a Week 12 visit and 75% of all subjects completing a Week 12 visit.

PK sampling collection for subjects to provide optional samples on Weeks 2 or 4, that were not able to provide optional PK samples on Day 1 was changed to: Optional sample collection on Day 1, Week 2, or Week 4 are not dependent on collection at any prior or subsequent sample collection time.

## 5.0 Study Objectives

## 5.1 Primary Objectives

The primary objective of the study is to evaluate the potential for ABI-H0731 to increase the rapidity of HBV DNA decline in hepatitis B "e" antigen (HBeAg) positive chronic hepatitis B infection (CHB) subjects by initiating treatment with ABI-H0731 + ETV in subjects who are not yet on treatment for CHB, as measured by timing and magnitude of change in serum HBV DNA from Baseline.

PRS 005 T 17 G 


#### 5.2 Secondary Objectives

The following secondary objectives are defined for this study:

- To evaluate the safety and tolerability of ABI-H0731 in combination with ETV therapy as initial therapy for HBeAg-positive CHB subjects.
- To confirm a lack of drug-drug interactions between ETV and ABI H0731.
- To evaluate the potential for emergence of resistance, if any, for ABI-H0731 in combination with ETV therapy.

#### 5.3 Exploratory Objectives

The following exploratory objectives are defined for this study:

- To evaluate the kinetics of and absolute changes from Baseline in biomarkers of transcriptionally active cccDNA (HBeAg and HBsAg)
- To evaluate the kinetics of and absolute changes from Baseline in circulating hepatitis B virus (HBV) RNA
- To assess the relationship between changes in exploratory viral biomarkers such as changes in viral RNA and hepatitis B core-related antigen (HBCrAg) with clinical outcomes
- To explore the pharmacokinetics (PK) of ABI-H0731
- For subjects who provide an optional pharmacogenomic (PG) sample, to evaluate the potential contribution of host genomics to outcomes

## 6.0 Study Design

This Phase 2a, multi-center, randomized, double-blind, placebo-controlled study will assess the safety, efficacy, PK, and pharmacodynamics of 300 mg ABI-H0731 daily in combination with ETV in treatment-naïve subjects with HBeAg-positive CHB. Twenty-four subjects will be randomized in a 1:1 ratio to receive investigational agent (ABI-H0731 or matching placebo) as add-on therapy to ETV for up to 6 months. ETV will continue uninterrupted for the duration of the study as well as during follow-up.

Safety will be monitored by a Data Monitoring Committee (DMC) when approximately 25% and 75% subjects (across ASM31201-731201 Amendment 3 v4.0 / 09 November 2018 and ASM31202-731202 studies Amendment 1 v2.1 / 30 July 2018 [UK only] Amendment 1 v2.0 / 18 June 2018 [USA, Canada, NZ, HKG] studies) complete their Week 12 visit (or discontinued study without completing Week 12). This timing differs from that defined in the protocol, to allow for earlier identification of potential safety concerns. There will be an assessment of PK data after all subjects have completed Week 4 (or discontinued study without completing Week 4) to confirm a lack of an important impact of ABI-H0731 on the steady-state PK of ETV.

At the end of the 24-week treatment period in this study, subjects will either continue ETV and stop treatment with ABI-H0731/placebo, or they may elect to roll over onto the optional, open-label, extension study ABI-H0731-211.

Subjects who do not roll into optional open-label study ABI-H0731-211 will continue on ETV alone and will be monitored for an additional 12 weeks to determine if any changes in either viral antigens or viral RNA which may have been noted on treatment will persist through end of follow-up.

Subjects who do elect to roll over to the optional, open-label, extension study of ABI-H0731 + SOC NUC (protocol ABI H0731-211) will continue on open-label combination therapy as per that study. The objective of the extension study, ABI-H0731-211, will be to evaluate the safety and potential for benefits of up to one additional year of therapy with ABI-H0731 in combination with SOC NUC therapy. Subjects will be required to sign a separate informed consent form prior to entering the ABI H0731-211 study.

PRS 005 T 17 G 


#### 6.1 Sample Size Considerations

As a proof-of-concept trial, there are no statistical hypotheses, per se, regarding treatment effects in this study. Rather, displays and comparisons of study results, regarding dose-related safety, efficacy, and PK profiles among the treatment groups, will primarily utilize descriptive statistics.

The primary objective of the study will be measured by changes from Baseline to Week 12 or Week 24 in mean log<sub>10</sub> HBV DNA. As the results for this study will be used to collect information for future studies, both timepoints will be reviewed independently, with no control of the alpha level.

With a sample size of 24 subjects, randomized in a 1:1 ratio (12 ABI-H0731:12 placebo), a 2-sample t-test for mean difference with a 2-sided 0.05 significance level has 87.7% power to detect a difference of at least 0.4 log<sub>10</sub> (IU/mL) in the change from Baseline in serum HBV DNA level at Week 12 or Week 24 between the placebo + ETV and ABI-H0731 + ETV groups, where an equal standard deviation of 0.3 is assumed for both groups (Table 1).

Table 1 Power Calculations under Various Mean Differences in the Change from Baseline in HBV DNA levels at Week 12 or 24 between Treatment Groups

| Estimated mean difference at Week 12 or Week 24 between placebo + ETV and | Power for N=24 subjects<br>(12 ABI-H0731 + ETV: 12 Placebo + ETV) | | | |
|---|---|---|---|---|
| ABI-H0731 + ETV groups Change from<br>Baseline HBV DNA levels | SD = 0.25 | SD = 0.30 | SD = 0.50 | SD = 0.60 |
| 0.25 log <sub>10</sub> IU/mL | 0.649 | 0.497 | 0.216 | 0.164 |
| 0.30 log <sub>10</sub> IU/mL | 0.802 | 0.649 | 0.290 | 0.216 |
| 0.40 log <sub>10</sub> lU/mL | 0.963 | 0.877 | 0.466 | 0.346 |
| 0.50 log <sub>10</sub> IU/mL | 0.997 | 0.974 | 0.649 | 0.497 |
| 0.60 log <sub>10</sub> IU/mL | >0.999 | 0.997 | 0.802 | 0.649 |

Calculated using SAS, based on a two-sided, two-sample t-test for mean differences, assuming equal weight of treatment groups, and alpha=0.05. ETV=entecavir; HBV=hepatitis B virus; SD=standard deviation.

#### 6.2 Randomization

Approximately twenty-four subjects will be randomized in a 1:1 ratio (12 ABI-H0731:12 placebo) by an independent Interactive Web Response System (IWRS) vendor.

#### 6.3 Schedule of Assessments

The study schedule of assessments per Amendment 1 v2.1 dated 30-July-2018 is noted in Table 2.

PRS 005 T 17 G 



Statistical Analysis Plan


#### **Table 2. Schedule of Assessments**

| Period or Visit | Screening | | | | On Tre | atment | | | | Fallo | w-Up <sup>a</sup> | Premature<br>Termination <sup>b</sup> | Unscheduled <sup>c</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day or Week | Day (-45) to<br>Day (-1) | Day 1 | Week<br>2 | Week<br>4 | Week<br>8 | Week<br>12 | Week<br>16 | Week<br>20 | Week<br>24 a | Week<br>28 | Week<br>36 | Varies | Varies |
| • | indow (days) | 0 | +/- 2 | +/- 2 | +/- 3 | +/- 3 | +/- 3 | +/- 3 | - 3 | +/- 3 | +/- 3 | N/A | N/A |
| Informed Consent(s) d | X | Ů | | | | | | | X <sup>1</sup> | ., 5 | | 1,111 | 1011 |
| Demographic data | X | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | |
| Medication history | X | | | | | | | | | | | | |
| Liver screening e | X | | | | | | | | | | | | |
| Full physical examination | X | | | | | | | | X | | X | X | |
| 12 Lead ECG | X | X | | | | X | | | X | | X | X | if indicated |
| Height and weight | X | X | | X | | | | | X | | X | | |
| Vital signs | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medications /<br>Adverse events | | X | X | X | X | X | X | X | X | X | X | X | X |
| Confirm eligibility | | X | | | | | | | | | | | |
| Randomization (IRT) | | X | | | | | | | | | | | |
| Symptom directed physical exam <sup>m</sup> | | X | X | X | X | X | X | X | | X | | | X |
| Paper diary | | X | X | X | X | X | X | X | X | | | | |
| Drug accountability | | | X | X | X | X | X | X | X | X | $\mathbf{X}^{\mathrm{j}}$ | if applicable | |
| Drug dispensation | | X | X | X | X | X | X | X | X | $X^{j}$ | | | |
| In-clinic dosing:<br>ABI-H0731/placebo | | X | X | X | X | X | X | X | X | | | | |
| ETV dosing <sup>k</sup> | | $X^k$ | $X^k$ | $X^k$ | X | X | X | X | X | X | | | |
| Digital photography <sup>c</sup> | | | | | | | | | | | | | if indicated |
| Virology/Immunology | | | | | | | | | | | | | |
| HBV genotype | X | | | | | | | | | | | | |
| HBV viral load | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Quant HBsAg, quant<br>HBeAg <sup>f</sup> | X | X | | X | X | X | X | X | X | X | X | X | X |
| HBsAb, HBeAb | X | X | | | | X | | | X | | X | X | |
| HBV RNA | X | X | X | X | X | X | X | X | X | X | X | X | X |



Statistical Analysis Plan


| | Period or Visit | Screening | | | | On Tre | atment | | | | Fallo | w-Up <sup>a</sup> | Premature Termination <sup>b</sup> | Unscheduled <sup>c</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| s | Study Day or Week | Day (-45) to<br>Day (-1) | Day 1 | Week<br>2 | Week<br>4 | Week<br>8 | Week<br>12 | Week<br>16 | Week<br>20 | Week<br>24 a | Week<br>28 | Week<br>36 | Varies | Varies |
| HBV DNA | serum resistance | | X | X | X | X | X | X | X | X | X | X | X | X |
| HIV Ab | | X | | | | | | | | | | | | |
| HCV Ab; H<br>(IgM); HEV | HDV Ab; HAV<br>V (IgM) | X | | | | | | | | | | | | X |
| Laboratory A | Assessment | | | | | | | | | | | | | |
| Chemistry <sup>b</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematolog | y | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Coagulation | n | X | X | | X | X | X | X | X | X | X | X | X | X |
| Serum AFP | ) | X | | | | | | | | | | | | |
| FSH (femal | les only) | X | | | | | | | | | | | | |
| Urinalysis | | X | X | | X | X | X | X | X | X | X | X | X | X |
| Urine drug | test | X | X | | | | | | | | | | X | X |
| Pregnancy ' | Test <sup>g</sup> | X | X | X | X | X | X | X | X | X | X | | X | X |
| PK Sample | Collection | | | | | | | | | | | | | |
| Pre-dose h | ABI-H0731 | | X | X | X | | X | | | X | X | | X | X |
| Pre-dose " | ETV | | X | X | X | | X | | | X | X | | X | X |
| Optional po<br>4 (±2) hour<br>H0731 and<br>administrat | rs after ABI-<br>ETV | | X | X | X | | | | | | | | | |
| Exploratory | | | | | | | | | | | | | | |
| Optional PG | sample <sup>c</sup> | | X | | | | | | | | | | | |
| Core protein | (HBCrAg) | | X | X | X | X | X | X | X | X | X | X | X | X |
| Viral nucleic | | 11 . 1 . | X | X | X | X | X | X | X | X | X | X 1.6 | X | X |

a Subjects who elect NOT to enter rollover study ABI-H0731-211 at Week 24 will discontinue ABI-H0731 and continue to take ETV during the 12-week follow-up period (inclusive of Weeks 28 and 36).

physical examination and the following laboratory tests: ALT, AST, total bilirubin, INR, and serum albumin. If the ALT flare is confirmed, perform the following tests: HBV DNA, quantitative HBV serologies (quantitative HBeAg [reflex qualitative HBeAg if quantitative HBeAg is negative]), HAV IgM, HCV RNA, HDV RNA, and HEV IgM

b Subjects who discontinue treatment before Week 24 should immediately undergo the assessments listed for the Premature Termination visit and then continue scheduled assessments, except that these subjects need only two further PK collections (at the Premature Termination visit and the next scheduled time point). Subjects who discontinue study assessments before completing the 12-week follow-up period should undergo the assessments listed for the Premature Termination visit.

c Any subjects with rash or ALT flare (defined as ALT≥2×Baseline and ≥10×ULN) should return to the clinic for an unscheduled visit as soon as possible, ideally within 3 days.

Unscheduled visit for ALT flare: All subjects should have the laboratory findings confirmed within 3 days of receipt of the original results. All subjects should undergo a symptom directed



Statistical Analysis Plan


Unscheduled visit for rash: Digital photographs of the rash should be taken and blood samples should be taken (for erythrocyte sedimentation rate, complete blood count [with differential], creatinine, ALT, AST, and total bilirubin). If the rash diagnosis is uncertain, or if a rash is Grade 2, a referral to a dermatologist should be made and a biopsy should be conducted if recommended by the dermatologist. For a rash that is Grade 3 or higher, a referral to a dermatologist should be made and a biopsy should be requested of the dermatologist. All dermatologist reports and biopsy results will be included in the source and eCRF. Digital photographs of the rash should be obtained at each visit to document any change in condition. Unscheduled visits should continue until the rash has resolved or declined to Grade 1 or less for two successive visits.

- d Study specific including optional PG consent. PG sample collection requires documentation of completed PG consent.
- Liver evaluation to be done by any protocol approved method (Biopsy, fasting FibroScan, MRI, liver ultrasound), unless a liver biopsy demonstrating lack of cirrhosis or bridging fibrosis has been conducted in the last 6 months.
- f If quantitative HBsAg or HBeAg are negative at any visit subsequent to Screening, reflex to qualitative.
- g A serum pregnancy test is required at screening, and on Day 1 both urine and serum should be performed (subjects may begin treatment based on urine results; any subjects negative by urine subsequently found to be positive on serum should immediately discontinue treatment and may be replaced). All post-Day 1 pregnancy tests may be conducted by urine dipstick. If positive on dipstick, please reflex to serum.
- h If the subject inadvertently administers study drug prior to collection, a PK sample should still be drawn. Refer to the protocol PK Assessments section.
- i Optional post-dose PK samples for ABI-H0731 and ETV may be collected 4 (±2) hours after in-clinic study drug + ETV administration at Day 1 and either Week 2 or Week 4. If a subject can only provide optional samples on Weeks 2 or 4, then those may be collected from subjects that were not able to provide optional PK samples on Day 1.
- j Week 28 drug dispensation and Week 36 drug accountability only applies to ETV, not to ABI-H0731/placebo.
- k If subjects are not able to remain in clinic for ETV dosing, then ETV may be dosed following their clinic visit and subjects should be reminded to record the dosing time within their dosing diary.
- 1 Subjects who elect to roll over onto the open-label extension study will be required to sign a separate consent at Week 24.
- m Dermatology assessments were added based on protocol v2.1 for UK only.

Ab=antibody; AFP=alfa fetoprotein; ALT=alanine aminotransferase; AST=aspartate aminotransferase; ECG=electrocardiogram; eCRF=electronic case report form; ETV=entecavir; FSH=follicle-stimulating hormone; HAV=hepatitis A virus; HBCrAg =hepatitis B core-related antigen; HBeAb=HBeAg antibody; HBeAg=hepatitis B "e" antigen; HBSAb=HBsAg antibody; HBsAg=hepatitis B surface antigen; HBV=hepatitis B virus; HCV=hepatitis C virus; HDV=hepatitis D virus; HEV=hepatitis E virus; HIV=human immunodeficiency virus; IgM=immunoglobulin M; MRI=magnetic resonance imaging; N/A=not applicable; PG=pharmacogenomic; PK=pharmacokinetic; Quant=quantitative; ULN =upper limit of normal.

Statistical Analysis Plan


## 7.0 Study Endpoints, Variables and Covariates

#### 7.1 Efficacy Endpoints and Variables

#### 7.1.1 Primary Efficacy Endpoints

The primary efficacy endpoint is two co-primary endpoints:

- 1) the mean change from baseline in log<sub>10</sub> HBV DNA at Week 12
- 2) the mean change from baseline in log<sub>10</sub> HBV DNA at Week 24

using a HBV DNA transfection-based assays against representative HBV strains of genotypes A, B, C, and D

#### 7.1.2 Secondary Endpoints

The primary efficacy variable, HBV DNA, will be collected at Screening, Day 1, and Weeks 2, 4, 8, 12, 16, 20, and 24 (or at the time of discontinuation)

Follow-up samples will be collected Weeks 28 and 36 for subjects who do not continue treatment in the extension protocol (ABI-H0731-211). Subjects who enter the ABI-H0731-211 protocol will have samples collected according to that protocol.

The following secondary endpoints will be evaluated using these variables:

- Percent of subjects with a decline in viral DNA to below limit of quantitation (LOQ) at end of treatment
- Median time to viral suppression, defined as HBV DNA <20 IU/mL</li>
- Incidence of Emergence of resistant HBV variants, if any

Other Secondary Endpoints include:

- Drug concentrations:
  - o Trough levels and (in subjects where optional samples are available) trough to peak ratios of ABI-H0731 on ABI-H0731 + ETV
  - o Trough levels and (in subjects where optional samples are available) trough to peak ratios of ETV on ABI-H0731 + ETV therapy as compared with placebo + ETV

Safety endpoints as outlined in Section 7.2 will be evaluated.

#### 7.1.3 Exploratory Efficacy Endpoints

Blood samples for the assessment of secondary and exploratory efficacy endpoints are collected according to the Schedule of Assessments (Table 2). These assessments include HBV DNA, quantitative/qualitative HBsAg and HBeAg levels, HBsAg antibody (HBsAb) and HBeAg antibody (HBeAb), HBV RNA, HBCrAg, and HBV resistance samples.

Follow-up samples will be collected at Weeks 28 and 36 for subjects who do not continue treatment in the extension protocol. Subjects who enter the optional extension protocol (ABI-H0731-211) will have samples collected according to that protocol.

Reporting for assessments of HBeAg seroconversion (loss) will include only those subjects with detectable (positive) HBeAg viral antigen at baseline.

Reporting for assessments of HBV RNA will include only those subjects with detectable (positive) HBV RNA at baseline.

Statistical Analysis Plan


The assessments will be reported using Covance labs, or Assembly Labs. The incidence of LOQ values for each of these assessments will be reported and for numerical summaries the value at LOQ will be reported.

The following exploratory endpoints will be evaluated using these variables:

- The mean change from baseline in serum viral antigen (HBsAg, HBeAg, and HBCrAg) levels at each time point where collected
- Percent of subjects with loss (defined as below LOQ) or decline in HBsAg or HBeAg (<0.5 log<sub>10</sub>, ≥0.5 to 1.0 log<sub>10</sub>, or >1.0 log<sub>10</sub> decrease in viral antigen) at end of treatment (Week 24)
- Percent of subjects with HBsAg seroconversion (loss of HBsAg and appearance of HBs antibody) or HBeAg seroconversion (loss of HBeAg and appearance of HBe antibody) at each timepoint
- Change from Baseline in mean log<sub>10</sub> viral RNA at each timepoint
- Percent of subjects whose HBV DNA achieves "target not detected" at each timepoint
- For subjects who do NOT rollover onto the optional extension study, ABI-H0731-211:
  - Percent of subjects with suppression of detectable serum HBV RNA on treatment whose HBV RNA rebounds after discontinuing treatment during Post-Treatment follow-up with ABI-H0731 + ETV as compared with placebo + ETV
  - Percent of subjects with changes in HBsAg or HBeAg whose viral antigen rebounds after discontinuing treatment during Post-Treatment follow-up with ABI-H0731 + ETV as compared with placebo + ETV
  - Percent of subjects with HBsAg or HBeAg loss at Week 24 that is maintained through the end of Post-Treatment follow-up (Week 36) after discontinuing treatment with ABI-H0731 + ETV as compared with placebo + ETV

HBV resistance testing, using exploratory research samples, will be performed on subjects with evidence of nonresponse to treatment, to assess potential HBV core gene sequences associated with viral resistance or blunted treatment response, viral DNA rebound (>1 log10 HBV DNA rebound from on treatment nadir) or viral load plateauing (≥2 consecutive samples with viral load remaining within 0.5 log10 of nadir).

Pharmacogenomic samples will be collected at Day 1 for subjects who consent to this procedure. These samples may be saved for future research. If differences are noted in outcomes between racial or ethnic groups, the correlation between PG variables with clinical outcomes may be evaluated for subjects who provide optional informed consent.

## 7.2 Safety Endpoints and Variables

The safety variables noted in this section will be used to evaluate the following set of secondary safety endpoints:

- Number of subjects with adverse events (AEs), premature discontinuations, abnormal safety laboratory results, electrocardiogram (ECG), or vital signs
- Subjects with abnormal alanine aminotransferase (ALT) at Baseline who have normal ALT at Week 24 on ABI-H0731 + ETV therapy as compared with placebo + ETV therapy

#### 7.2.1 Adverse Events

Adverse events will be coded using MedDRA 21.0 (March 2018) and graded by Medidata Rave Coding tool. Adverse events will be monitored and reported from the time written informed consent is signed until completion of the Week 36 follow-up visit or until 30 days following cessation of the last dose of treatment with the study drug for subjects who discontinue from follow-up.

Statistical Analysis Plan


An AE is defined as any untoward medical occurrence in a study subject administered an investigational product(s) regardless of the causal relationship with treatment.

An AE, therefore, can be any unfavorable and unintended sign (including laboratory finding), symptom, or disease temporally associated with participation in an investigational study, whether or not considered drug related. In addition to new events, any increase in the severity or frequency of a pre-existing condition that occurs after the subject signs the Informed Consent Form (ICF) for participation is considered an AE. This includes any side effect, injury, toxicity, or sensitivity reaction.

An AE will be considered a Treatment-emergent AE (TEAE) if it first occurs or begins previous to and worsens on or after the first study drug dose date and before the last dose date + 30 days.

The following AE details will be recorded on the eCRFs:

- Adverse event (verbatim)
- Whether the AE is an adverse event of special interest (AESI). AESI's include rash and ALT flare.
- Start / end date of the AE
- Whether the AE is serious or not, and if yes, which category (AE resulted in death; AE is life-threatening; AE resulted in persistent or significant disability or incapacity; AE resulted in initial or prolonged hospitalization; AE is associated with a congenital anomaly or birth defect; AE is a medically important event not covered by other criteria).
- Relationship to Study Treatment (Not related; Unlikely related; Possibly related; Related)
- Action taken with Study Treatment (Dose not changed; Drug interrupted; Drug withdrawn; Not applicable; Unknown)
- Intensity (Mild (Grade 1); Moderate (Grade 2); Severe (Grade 3); Life threatening (Grade 4))
- Outcome (Fatal; Not recovered/not resolved; Recovered/resolved; Recovered/resolved with sequelae; Recovered/resolving; Unknown)
- Non-study drug treatment received for the AE

The intensity of each AE and laboratory abnormality will be assessed by the Investigator according to the modified Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (noted in APPENDIX II of the protocol), which grades the severity of clinical AEs and laboratory abnormalities in a four-category system.

#### 7.2.2 Clinical Laboratory Tests

Clinical laboratory tests will be performed at the timepoints indicated in the Schedule of Assessments (<u>Table 2</u>). The clinical laboratory assessments are listed in <u>Table 3</u>.

PRS 005 T 17 G 



Statistical Analysis Plan


#### Table 3 Clinical Laboratory Tests

| Panel | Tests |
|---|---|
| Clinical chemistries | Blood glucose levels, serum or plasma electrolytes (sodium, potassium, chloride, bicarbonate), calcium, blood urea nitrogen, creatinine, uric acid, total and direct bilirubin a, ALT, AST, GGT, alkaline phosphatase, LDH, amylase, triglycerides, total cholesterol, inorganic phosphate or total phosphate, total protein, albumin, lipase, and total serum or plasma globulins |
| In case of ALT flares | ALT, AST, total bilirubin, serum albumin, and INR |
| Hematology | Complete blood counts: hemoglobin, hematocrit, RBC indices (MCV, MCHC), reticulocyte counts, leukocyte counts (total and differential), and platelet counts |
| Coagulation | Prothrombin time, INR and aPTT |
| Urinalysis | pH, specific gravity, protein, glucose, ketones, and occult blood |
| Other | AFP, HbA1c, and FSH |
| Pregnancy tests | For females only; a serum or plasma pregnancy test must be performed at screening, and both serum/plasma and urine are required Day 1; a serum, plasma, or urine pregnancy test must be performed at all subsequent visits. A positive result disqualifies the subject for study treatment |
| Urine drug<br>screening | Amphetamine/methamphetamine, barbiturates, benzodiazepines, cannabinoids, cocaine metabolite, ecstasy, ethanol, opiates, phencyclidine, and propoxyphene. Note: If cannabinoids are not illegal in the subject's local, cannabinoids are not exclusionary |
| Antibodies | HCV, HDV, HAV IgM, HEV IgM, and HIV |

AFP=alpha fetoprotein; ALT=alanine aminotransferase; aPTT=activated partial thromboplastin time; AST=aspartate aminotransferase; FSH=follicle-stimulating hormone; GGT=gamma-glutamyl transpeptidase; HAV=hepatitis A virus; HbA1c=hemoglobin A1c; HCV=hepatitis C virus; HDV=hepatitis D virus; HEV=hepatitis E virus; HIV=human immunodeficiency virus; IgM=immunoglobulin M; INR=International Normalized Ratio; LDH=lactate dehydrogenase; MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume; RBC=red blood cell; ULN=upper limit of normal

a Perform fractionated bilirubin, if total bilirubin >ULN.

During the study, any clinically significant laboratory abnormality or clinically significant change from Baseline will be recorded as an AE.

#### 7.2.3 Vital Signs

Vital signs will be collected at Screening, Day 1, and Weeks 2, 4, 8, 12, 16, 20, and 24 (or at the time of discontinuation). Follow-up samples will be collected Weeks 28 and 36 for subjects who do not continue treatment in the extension protocol.

Variables will include temperature, systolic blood pressure, diastolic blood pressure, pulse rate, and respiratory rate. Additionally, height, weight, and body mass index (BMI) will be collected on the CRF at screening, with weight collected again at Day 1, and Weeks 4 and 24, and Week 36 for subjects who remain in the follow-up period.

#### 7.2.4 12-Lead ECG

Twelve-lead ECG will be collected at screening, Day 1, and Weeks 12, and 24 (or at the time of discontinuation). Follow-up samples will be collected at Week 36 for subjects who do not continue treatment in the extension protocol. During the study, any clinically significant ECG result should be confirmed, and if confirmed, should be recorded as an AE.

PRS 005 T 17 G 


#### 7.3 Pharmacokinetic Endpoints and Variables

The pharmacokinetic endpoints for this study are as follows:

- Trough levels and (in subjects where optional post-dose samples are available) trough to peak ratios of ABI-H0731 on ABI-H0731 + ETV therapy
- Trough levels and (in subjects where optional post-dose samples are available) trough to peak ratios of ETV on ABI-H0731 + ETV therapy as compared with placebo + ETV therapy

Pre-dose drug concentration samples will be collected to determine trough concentrations of ABI-H0731 and ETV. Post-dose samples for both ABI-H0731 and ETV will be collected from subjects willing and able to provide the sample  $4 \pm 2$  hours after in-clinic dosing. Sample timing is outlined in <u>Table 4</u>.

Table 4: Pharmacokinetic Sample Collection

| Time Period | Timepoint <sup>a</sup> | Time Relative to Study Drug Administration <sup>b</sup> |
|---|---|---|
| | Study Day 1 pre-dose | Before |
| Double-Blind | Study Weeks 2, 4, 12, 24 pre-dose | Before |
| Treatment | OPTIONAL ° | 4 (±2) hours post-dose |
| | Day 1, Week 2, and/or Week 4, post-dose (see laboratory manual) | |
| Follow-Up | Study Week 28 pre-dose <sup>e</sup> | Collect at same time with other central labs |

a A PK sample should be collected if an unscheduled or premature termination visit is performed.

- b Sample collection times are targeted times. Samples collected outside of these targeted times will not be considered protocol deviations as long as the actual time the sample is collected is accurately recorded on source documentation and the case report form.
- c If a subject can only provide optional samples on Weeks 2 or 4, those may be collected from subjects that were not able to provide optional PK samples on Day 1.

#### 7.4 Other Variables

Other assessments that will be collected and included for analyses include:

- Demographic characteristics, including sex, ethnicity and race
- Liver screening using Fibroscan categorization method of F0 through F2.
- Prior and concomitant medications
- HBV treatment history
- Medical and surgical history
- Procedures
- Complete and symptom-directed physical examinations
- Drugs of Abuse testing
- Pregnancy testing


Exposure and compliance to study medication

#### 7.5 Predetermined Covariates and Prognostic Factors

Race, ethnicity, and/or HBV genotype (A, B, C, D, E-H) may be used as a covariate where indicated within the analysis.

#### 8.0 **Definitions**

The following table will be used to define variables used within the statistical tables, figures, and listings.

Table 5 Variables and Definitions

| Variable | Definition |
|---|---|
| Baseline | Baseline is defined as the value closest to but prior to the initiation of study drug administration. |
| Change from baseline | Change from baseline will be defined as the post-baseline value minus the baseline value, where applicable (on a subject level). Change from baseline will only be calculated for subjects who have both baseline and at least one post-baseline value for any parameter. |
| Study day | Study Day 1 will be based on the date of first dose. Events prior to this day will be reported as a negative study day (i.e. there will be no Day 0). The study day of an event will be calculated as (event date) – (first dose date) when the event occurred prior to first dose, and (event date) – (first dose date) + 1 when the event occurred after first dose. |
| Duration Variables | Duration variables (ex. time in study, exposure to study drug treatment, days since last visit, duration of AEs, etc.) will be calculated using the general formulas below: |
| | Duration (days) = (End date - Start date) + 1 |
| | Duration (weeks) = Duration (days) / 7 |
| | Duration (months) = Duration (days) / 30.25 |
| Body Mass Index (BMI) | Where not collected on the eCRF, BMI will be calculated as: |
| | BMI = Weight (kg) / Height (m) <sup>2</sup> |

## 9.0 Analysis Sets

#### 9.1 Intent-to-Treat

The Intent-to-treat (ITT) population will be defined as all randomized subjects. Subjects in this population will be analyzed according to their randomized treatment assignment, regardless of the actual treatment received.

## 9.2 Safety

The safety population will include all randomized subjects who used any amount of study drug. Subjects in this population will be analyzed according to the actual treatment received.

PRS 005 T 17 G 


#### 9.3 Pharmacokinetic

Pharmacokinetic Population 1 (PK1): The PK1 population will include all subjects in the safety population who have ABI-H0731 PK data assessments available.

Pharmacokinetic Population 2 (PK2): The PK2 population will include all subjects in the safety population who have ETV PK data assessments available.

#### 9.4 Pharmacogenomic

The pharmacogenomic (PG) population will consist of subjects who have consented to, and have provided, an optional PG sample. Subjects in this population will be analyzed according to the actual treatment received.

## 10.0 Interim Analyses

No formal interim analyses are planned, however, there will be a Week 4 PK analysis as well as a Data Monitoring Committee (DMC) safety analyses for data collected to Week 12. The unblinded statistician and programmer will provide these analyses, as indicated in <u>Section 6.3</u>.

## 10.1 Week 4 Pharmacokinetic Analysis

After all subjects have completed Week 4 (or discontinued before completing Week 4), PK data will be reviewed by an unblinded pharmacology reviewer to verify whether ETV steady-state exposure are affected by combination treatment with ABI-H0731.

Results will be provided once and will include trough levels and trough to peak ratios (as available) for ABI-H0731 and ETV concentrations in tabular and graphical format.

These results will be provided for the PK1 and PK2 Populations in an unblinded manner by treatment group, delivered by the unblinded PRA statistician or by a PRA PK expert. The unblinded PK results will be posted on a user-restricted study portal to ensure that only the intended recipients have access to the results. The unblinded recipients will be notified of when results are posted to complete their review of the unblinded PK data.




| Name: Title and Company | Email: |
|-------------------------|--------|

#### 10.2 Week 12 Safety Analysis

A DMC external to the Sponsor and the CRO will be formed with members consisting of individuals chosen for their expertise in treatment of HBV. Members of the DMC will include, at a minimum, physicians external to the Sponsor and the CRO and appropriate statistical representation. The primary role of this independent DMC will be to monitor unblinded safety data.

Details of the DMC will be outlined separately in a DMC Charter. The DMC Charter will detail data to be analyzed, and will identify members of the DMC, responsibility of those members, and frequency of meetings.

These results will be provided to the DMC members and the Sponsor's designated unblinded statistician in an unblinded manner delivered by the unblinded PRA statistician for posting on a user-restricted study portal, to ensure that only the intended recipients have access to the results. The unblinded recipients will be notified when results are posted. Details of the distribution of data outputs to the DMC members and sponsor's designated unblinded statistician will be outlined in the DMC Charter.

The list of statistical outputs to be produced for the DMC members and the unblinded Sponsor statistician will be documented in the ABI-H0731-201 and 202 DMC Data Transfer Plan; including a separate set of unblinded TFL shells for unblinded DMC members and the unblinded Sponsor statistician and a separate set of blinded TFLs for the blinded Sponsor team members.

#### 11 0 Data Review

#### 11.1 Data Handling and Transfer

Details regarding the data handling, including how data is received by external vendors and which data is included in cleaning and transfers of data, are referenced in the project's Data Management Plan.

#### 11.2 Data Screening

Beyond the data screening built into the PRA Data Management Plan, the PRA programming of analysis datasets and TFLs provides additional data screening. Presumed data issues will be output into SAS logs identified by the word "Problem" and extracted from the logs by a SAS macro and sent to Data Management.

Review of a pre-freeze TFL run on clean subjects and a post-freeze TFL run on the frozen database allow for further data screening prior to lock. The post-freeze TFL will be discussed with the sponsor in a data review meeting to identify any final data issues and seek corrections prior to database lock. The PRA statistician and the sponsor must approve database lock.

#### 12.0 Statistical Methods

#### 12.1 General Considerations

All analyses will use SAS version 9.4 or higher. Results will be reported by treatment group, based on the following test and reference product categories:

• **ABI-H0731**: This group will include subjects receiving test product ABI-H0731 in addition to their ETV therapy.

Statistical Analysis Plan


Placebo: This group will include subjects receiving placebo (matching placebo to ABI-H0731 tablets) in addition to their ETV therapy

Sites will be pooled together for all analyses.

Adjustments for multiplicity will not be made since this is a proof-of concept study. Separate inferences will be drawn for assessment.

Unless otherwise noted, categorical variables will be summarized using counts and percentages. Percentages will be rounded to one decimal place, except 100% will be displayed without any decimal places and percentages will not be displayed for zero counts.

Continuous variables will be summarized using the number of observations (n), mean, standard deviation (SD), median, minimum and maximum. The minimum and maximum values will be displayed to the same level of precision as the raw data, the mean and median to a further decimal place and the SD to two additional decimal places.

Confidence intervals will be two-sided and use the Clopper-Pearson (exact binomial) method at a 95% confidence level.

#### 12.2 Handling of Missing Data / Imputation Methods

All attempts will be made to prevent missing data.

To assess robustness of the primary efficacy variables, sensitivity analysis with missing values imputed by MMRM Using Multiple imputation (MI) will be performed see <a href="Appendix 2">Appendix 2</a> for multiple imputation method. Isolated missing values will be imputed by Markov Chain Monte Carlo (SAS PROC MI, MCMC) first to make the missing pattern monotone and then imputed by monotone linear regression. SAS PROC MI and PROC MIXED will be used to obtain MMRM estimates of treatment difference. SAS PROC MIANALYZE will be used to combine estimates and to generate the average test statistics for hypothesis testing. The Missing at Random method will be used with the following parameters MAR — assume missing at random, number of imputation=100, seed= SEED11 (for MCMC) and SEED12 (for MONOTONE REG) for imputation.

Missing data will only be imputed for the co-primary endpoints.

Percent of subjects with missing visits, and total missing visits per lab assessment may be summarized for the primary, secondary, and exploratory endpoints to assess the effect on repeated measures analysis for these endpoints.

All missing and partial dates for adverse events will be queried for a value. If no value can be obtained, substitutions will be made as detailed in <u>Table 6</u>. These substitutions will be used in calculations, however, the actual value recorded on the eCRF will be presented in all listings.

PRS 005 T 17 G 

Statistical Analysis Plan


Table 6. Adverse Event Start/Stop Date Imputation Imputation Rules for Partial Dates (D = day, M = month, Y = year)

| Parameter | Missing | Additional Conditions | Imputation |
|---|---|---|---|
| Start date for AEs | D | M and Y same as M and Y of first dose of treatment | Date of first dose of treatment |
| | | M and/or Y not same as date of first dose of treatment | First day of month |
| | D and M | Y same as Y of first dose of treatment | Date of first dose of treatment |
| | D dild ivi | Y prior to Y of first dose of treatment but same as Y of screening date | Date of screening date |
| | D, M, Y | None - date completely missing | Date of first dose of treatment |
| Stop date for AEs | | M and Y same as M and Y of last dose of treatment | Date of last dose of treatment |
| D | | M and/or Y not same as date of last dose of treatment | Use last day of month (i.e D may take on values of 28, 29, 30, or 31, depending on month) |
| D and M | | Y same as Y of last dose of treatment | Date of last dose of treatment |
| | | Y not same as Y of last dose of treatment | Use Dec 31 |
| | D, M, Y | None - date completely missing | No imputation, but assume ongoing |

D=day, M=month, Y=year

Note: In all cases, if an estimated start date is after a complete stop date, use the first day of the stop date month. Similarly, if the estimated stop date is before a complete or imputed start date, use the last day of the start day month.

In all cases, if it cannot be determined if the AE occurred prior to or after the first dose of treatment, the AE should be defined as treatment emergent.

In the event that an AE has missing results for relationship to study treatment the AE will be assumed to be related. If intensity of AE is missing, then no imputation will be applied.


#### Table 6. Prior and Concomitant Medications Start/Stop Date Imputation

Imputation Rules for Partial Dates (D = day, M = month, Y = year)

| Parameter | Missing | Additional Conditions | Imputation |
|---|---|---|---|
| Start date for | ate for D only M and Y same as M and Y of first | | Date of first dose of study |
| con meds | | dose of study drug | drug |
| | | M and/or Y not same as date of first dose of study drug | First day of month |
| | M and D | Y same as Y of first dose of study | Date of first dose of study |
| | | drug | drug |
| | | Y not same as Y of first dose of study drug | Use Jan 01 of Y |
| | M, D, and Y | None - date completely missing | Day prior to date of first dose of study drug |
| Stop date for | Stop date for D only M and Y same as M and Y of last | | Date of last dose of study |
| con meds | con meds dose of study drug | | drug |
| | | M and/or Y not same as date of last dose of study drug | Last day of month |
| | M and D | Y same as Y of last dose of study | Date of last dose of study |
| | | drug | drug |
| | | Y not same as Y of last dose of study drug | Use Dec 31 of Y |
| | M, D, and Y | None - date completely missing and | Date of last dose of study |
| | | NOT ongoing | drug |

Note: In all cases, if an estimated start date is after a complete stop date, use the first day of the stop date month.

Similarly, if the estimated stop date is before a complete or imputed start date, use the last day of the start day month.

For laboratory data, if the reported value of a parameter cannot be used in a statistical summary table (e.g., a character string is reported for a parameter of the numerical type), a coded value will be appropriately determined and used in the statistical analyses. In general, a value or lower limit of normal range such as '< 10' or '≤ 5' will be treated as '10' or '5' respectively, and a value or upper limit of normal range such as '> 100' will be treated as '100'. However, the actual values as reported in the database will be presented in data listings.

## 12.3 Subject Disposition

The number of screened subjects, subjects randomized, and subjects within each of the analysis populations (ITT, Safety, PK1, PK2, and PG) will be summarized by treatment group, and enrollment by site will be tabulated for subjects randomized into the study.

A list of subjects who did not meet all inclusion/exclusion criteria, and which criteria were not met, will be presented.

The number and percentage of subjects completing the study drug treatment period (up to and including Week 24), as well as the completion status of the study will be presented for each treatment group in the ITT population. Reasons for discontinuation from the study, as recorded on the eCRF, will be summarized (number and percentage) by treatment group. A listing of all subjects' disposition from the Treatment Phase and at end of study will be presented, along with the primary reason for discontinuation, as applicable. Percent of subjects who entered study 211 will be summarized by treatment group.

The number and percentage of subjects at each study visit will also be presented, and descriptive statistics will be used to summarize the total time in study from randomization in weeks.

PRS 005 T 17 G 


All disposition data will be included within listings.

#### 12.4 Protocol Deviations

Per PRA processes, protocol deviations data will be entered into a Clinical Trials Management System (CTMS). The study team and the sponsor will conduct on-going reviews of the deviation data from CTMS and the resulting set of evaluable subjects.

Deviations will be categorized into general categories: inclusion/exclusion criteria not met, study drug deviation (including storage issues, subject unblinding), prohibited medication received, overdose/misuse, study procedures not done (efficacy and safety), out of visit window, etc. The study team will also categorize protocol deviations as important or not important. Final review of protocol deviations will be conducted and finalized prior to unblinding the database.

The number of subjects with at least one major protocol deviation and the number of subjects with at least one minor protocol deviation within each deviation category will be presented by treatment group for the ITT population. Major and minor protocol deviations are defined per the study Protocol Deviation Guidance document.

#### 12.5 Demographic and Baseline Characteristics

Demographics will be summarized for the ITT, and Safety populations, and will include sex, race, ethnicity, age (in years, at time of signing informed consent), categorical age (i.e. < 65 years,  $\geq$  65 years – < 75 years,  $\geq$  75 years), weight, height, BMI, HBV genotype (A, B, C, D, E-H) if available, pre-treatment ALT levels, and ETV therapy reported at time of randomization.

All medical/surgical history, including those ongoing at screening, will be summarized in the ITT population based on the number and percentage of subjects reporting each event, as coded per Medical Dictionary for Regulatory Activities (MedDRA) v21.0. Current medical history events, denoted as 'ongoing' on the CRF, will be reported in a separate table.

All demographic and baseline characteristics, including HBV history (i.e. infection and diagnosis dates), and results from the screening liver examination, will be provided within data listings.

#### 12.6 Treatments

#### 12.6.1 Prior and Concomitant Medications

Medications received prior to or concomitantly with study drug will be categorized by Anatomical Therapeutic Classification (ATC) level 4 and preferred medication name, according to the WHODRUG dictionary (Version 2018MAR01 DDE B3). The number and percentage of subjects using each medication will be displayed by treatment group in the ITT population. Subjects will be counted only once for an ATC class and preferred term.

If a medication has an end date which occurs prior to the first dose of study drug, then it will be summarized as a prior medication. In the case where the medication end date is partially complete (i.e. missing day or month), then the month and/or year information will be used to determine if the medication was taken prior to study drug dosing, as applicable.

If a medication has a start date which occurs prior to the first dose of study drug and end date is after the first dose of study drug then it will be summarized as a concomitant medication.

All other medications with a start date after the first dose of study drug will be summarized as concomitant medications .


#### 12.6.2 Procedures

Procedures will be recorded from 7 days prior to the informed consent date through to study completion. All procedures will be summarized in the ITT population based on the number and percentage of subjects reporting each procedure, as coded per MedDRA v21.0.

#### 12.6.3 Compliance and Exposure to Study Drug

The summaries for compliance and exposure to study drug by treatment group will be presented for the Safety population.

For extent of study drug exposure, the duration will be calculated from Day 1 to the date of last study drug administration collected on the End of Treatment CRF. The expected total duration of on-treatment therapy for all subjects is 24 weeks. The distribution of subjects by the total number of weeks on therapy (i.e. < 1 week, 1-< 4 weeks, 4-< 8weeks, 8-< 12weeks, 12-<1 6weeks, 16-< 20weeks, and >=20 weeks) will be presented as will descriptive statistics for the total duration of days on therapy. This duration will be calculated as defined in the Section 8 Definitions.

In order to assess compliance with scheduled study drug dosing in the 24-week treatment period, the drug dispensing and return information collected on the drug accountability Case Report Forms will be used. Per protocol, each subject is expected to take three 100mg tablets every day during the treatment phase. In a 24-week period, a total of 504 tabs would be expected.

The percent compliance in 24 weeks will be calculated as:

% compliance = 100 \* 
$$\frac{Actual\ number\ of\ tablets\ taken}{Expected\ number\ of\ tablets\ over\ 24\ weeks}$$

where the actual number of tablets taken will be calculated as the *sum of all tablets dispensed* minus the *sum of all tablets returned* as reported on the Study Drug Accountability CRF, plus the number of tablets taken at each of the in-clinic dosing visits as reported in the Study Drug Administration CRF on Day 1, and Weeks 2, 4, 12, and 24. The expected number of tablets over 24 weeks is 504 or (last date subject took study drug – start date subject took study drug) + 1 as days exposed multiplied by 3 tablets daily.

Descriptive statistics for treatment compliance and the number and percentage of subjects at least 80% compliant will be presented by treatment group.

## 12.7 Efficacy Analyses

Summary statistics will be presented in the ITT, unless otherwise noted. For virology samples, a listing will be provided for the Safety population, and will include the following variables: HBV DNA (IU/mL), HBsAg (IU/mL), HBsAg (qualitative), HBeAg (IU/mL), HBeAg (qualitative), HBCrAg (IU/mL, and HBV RNA (copies/mL).

#### 12.7.1 Primary Endpoint Assessment: HBV DNA Change from Baseline

The primary endpoint is the mean change from baseline in log<sub>10</sub> HBV DNA at Week 12 and at Week 24.

The primary efficacy variable, HBV DNA, is collected at screening, Day 1, and Weeks 2, 4, 8, 12, 16, 20, and 24 (or at the time of discontinuation). Summary statistics will be provided by treatment group for the observed and change from baseline  $log_{10}$  serum results at the above study visits. Summaries will be provided for subjects in the ITT population. Mean change from baseline and 95% confidence intervals will be presented.

A repeated measures analysis using observed data from all scheduled visits for change from baseline in HBV DNA will be performed on the ITT population. This analysis will compare treatment groups over time using a linear mixed effects repeated measure model which includes fixed effects for treatment, visit, treatment-by-visit interaction, baseline value, baseline-by-visit interaction, and baseline covariates (baseline ALT, HBV genotype, time on historical HBV treatment). Unstructured covariance matrix will be

Statistical Analysis Plan


used. If there are convergence issues, then the use of first-order autoregressive (AR1) and/or the compound symmetry (CS) covariance matrices will be considered. The difference in least squares means between treatment groups and 95% confidence interval will be presented.

As this is a proof-of concept study, both primary timepoints of interest, Week 12 and Week 24 will be reviewed independently. There is no plan to control for alpha for reviewed timepoint, however, a significant difference at either timepoint would be considered clinically desirable and may warrant further exploratory investigation.

Graphs will be used to illustrate the changes from baseline for all post-baseline results up to Week 24. Results from both treatment groups will be presented on the same graph.

#### 12.7.2 Secondary and Exploratory Assessments

#### 12.7.2.1 ALT

For ALT Percent of subjects with normal value (within normal ranges as specified by central lab) at baseline and percent of subjects who continue to have normal ALT values at Week 24 will be provided by treatment group in the ITT population.

#### 12.7.2.2 HBV DNA Loss and Time to Viral Suppression

At each post-baseline timepoint, the number and percentage of subjects with detectable (>=LOQ) vs undetectable (<LLOQ) HBV DNA will be tabulated in the ITT population for each treatment group.

Time to viral suppression, defined as HBV DNA < 20 IU/mL, will be evaluated using Kaplan-Meier estimates for each treatment group. The summary will be provided based on results observed up to Week 24. A subject will be identified as having viral suppression if a HBV DNA of <20 IU/mL is observed for the subject, and all subsequent HBV DNA measurements are <20 IU/mL or below LOQ. Subjects will be considered censored for the Kaplan-Meier analysis if any of the following occur: 1) Subjects who are not observed to have encountered viral suppression by Week 24 (HBV DNA of <20 IU/mL) will be censored at their last observed visit up to week 24, 2) If a subject rebounds within the 24-week period, HBV DNA of <20 IU/mL occurs prior to Week 24 but a later assessment (HBV DNA of >=20 IU/mL) occurs then the overall status for that subject will be considered as censored at the first occurrence of a rebound, 3) if a subject discontinues study participation prior to an occurrence of HBV DNA of <20 IU/mL). The 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup> percentiles for time to viral suppression in weeks will be reported, along with the corresponding 95% confidence interval. An unstratified log-rank test will be used to assess differences in viral suppression rates between treatment groups.

#### 12.7.2.3 HBsAg, HBeAg, and HBCrAg levels

For HBsAg, HBcRAg, variables, summary statistics will be provided by treatment group for the observed and change from baseline  $\log_{10}$  serum results at each study visit. Summaries will be provided in the .ITT population. Mean change from baseline and 95% confidence intervals will be presented.

A repeated measures analysis using observed data from all scheduled visits for change from baseline in HBsAg, HBeAg, AND HBCRAg will be performed on the ITT population. This analysis will compare treatment groups over time using a linear mixed effects repeated measure model which includes fixed effects for treatment, visit, treatment-by-visit interaction, baseline value, baseline-by-visit interaction, and baseline covariates (baseline ALT, HBV genotype, time on historical HBV treatment). Unstructured covariance matrix will be used. If there are convergence issues, then the use of first-order autoregressive (AR1) and/or the compound symmetry (CS) covariance matrices will be considered. The difference in least squares means between treatment groups and 95% confidence interval will be presented.

PRS 005 T 17 G 




#### 12.7.2.4 HBsAg and HBeAg loss and seroconversion

The number and percentage of subjects with loss (defined as below LOQ) or decline in HBsAg or HBeAg (<0.5  $\log_{10}$ ,  $\geq$ 0.5 to 1.0  $\log_{10}$ , or >1.0  $\log_{10}$  decrease in viral antigen) will be tabulated for all measured visits in the ITT population. For HBeAg, the analytical measurement range is 0.11 –700.00 IU/mL. Samples with HBeAg concentrations greater than 700.00 IU/mL are diluted up to 1:2, extending the upper reporting limit to 1400.00 IU/mL. For HBsAg, the reportable range for the HBsAg quantitative assay is 0.05 – 124925.00 IU/mL. The analytical measurement range is 0.05 – 250.00 IU/mL. Samples with HBsAg concentrations greater than 250.00 IU/mL are diluted up to a maximum dilution of 1:500, extending the upper reporting limit to 124925.00 IU/mL.

Time to HBsAg loss and HBeAg loss will be evaluated using Kaplan-Meier estimates for each treatment group. The summary will be provided based on results observed up to Week 24. A subject will be identified as having loss if a result of <LOQ is noted for the subject, and all later records are <LOQ. Subjects will be considered censored for the Kaplan-Meier analysis if any of the following occur: 1) Subjects who are not observed to have HBsAg or HBeAg loss indicated by a result of <LOQ by Week 24 will be censored at their last observed visit up to week 24, 2) If a subject rebounds within the 24-week period, HBsAg or HBeAg < LOQ occurs prior to Week 24 but a later assessment of >=LOQ) occurs then the overall status for that subject will be considered as censored at the first occurrence of a rebound, 3) if a subject discontinues study participation prior to an occurrence of HBsAg or HBeAg < LOQ. The 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup> percentiles for time to loss in weeks will be reported, along with the corresponding 95% confidence interval. An unstratified log-rank test will be used to assess differences in loss rates between treatment groups.

Additionally, a Cox regression analysis will be used to determine association of the following baseline covariates on HBsAg and HBeAg loss: gender (male, female), race (Asian vs non-Asian), ethnicity (Hispanic/Latino, Non-Hispanic/Latino), and HBV genotype (A, B, C, D, E-H), as available. Hazard ratios and corresponding 95% Wald confidence limits will be provided in a summary table, along with the Wald Chi-Square p-value comparing the loss rates between the treatment groups.

Seroconversion status will be summarized at all post-baseline time points when antibodies for HBsAg and HBeAg are collected (i.e. Weeks 12, 24, and 36). For subjects where antibody is present, subjects with seroconversion will be presented as the number of subjects who also observed loss (i.e. HBsAg below LOQ, or HBeAg below LOQ) at the identified time point.

#### 12.7.2.5 HBV RNA

Summary statistics will be provided by treatment group for the observed and change from baseline log<sub>10</sub> viral RNA results at all study visits. Mean change from baseline and 95% confidence intervals will be presented.

A repeated measures analysis using observed data from all scheduled visits for change from baseline in HBV RNA will be performed on the ITT population. This analysis will compare treatment groups over time using a linear mixed effects repeated measure model which includes fixed effects for treatment, visit, treatment-by-visit interaction, baseline value, baseline-by-visit interaction, and baseline covariates (baseline ALT, HBV genotype, time on historical HBV treatment). Unstructured covariance matrix will be used. If there are convergence issues, then the use of first-order autoregressive (AR1) and/or the compound symmetry (CS) covariance matrices will be considered. The difference in least squares means between treatment groups and 95% confidence interval will be presented.

#### 12.7.2.6 Follow-up Subject Assessments

Follow-up efficacy assessments will be performed on ITT subjects who do not rollover onto the optional extension study, ABI-H0731-211.

For subjects with suppression of detectable serum HBV RNA (i.e. HBV RNA below LOQ) at Week 24, the number of subjects whose HBV RNA rebounds after discontinuing treatment will be presented at Weeks

PRS 005 T 17 G 


28 and 36 in both treatment groups. Similar analyses will be presented for both HBsAg and HBeAg for subjects with loss at Week 24, to determine whether results have rebounded following the treatment phase.

#### 12.7.2.7 Pharmacogenomic Assessments

Pharmacogenomic samples will be collected at Day 1 for subjects who consent to this procedure. These samples may be saved for future research. If differences are noted in outcomes between racial or ethnic groups from the Cox regression analysis defined in <u>Section 12.7.2.3</u>, the correlation between PG variables with clinical outcomes may be evaluated for subjects who provide optional informed consent.

A listing of PG results will be provided for the Safety population.

#### 12.8 Safety Analyses

#### 12.8.1 Adverse Events

Verbatim descriptions of AEs will be coded using Version 21.0 of MedDRA. Summary tables will be provided for all treatment-emergent adverse events (TEAEs) in the Safety Population.

A treatment-emergent AE is defined as any AE that newly appeared or worsened in severity on or after the first dose of study drug but not more than 30 days after the subject's last dose. If the start date of the AE is partial or missing, Table 5 in Section 12.2 will be used to determine the flag for treatment emergence.

An overall summary of TEAEs will be presented by treatment group and overall, and will include the following tabulations:

- the number of subjects reporting at least one TEAE, and the total the number of events reported
- the number of subjects with an Adverse Event of Special Interest (AESI) (i.e. ALT flare, rash, or other)
- the number of subjects with a treatment-related TEAE (i.e. either Possibly Related or Related)
- the number of subjects with Grade ≥3 (severe) TEAE
- the number subjects discontinuing the study due to a TEAE
- the number of subjects with at least one serious TEAE
- the number of subjects with a TEAE resulting in death.

Additionally, AEs will also be summarized as categorized by body system and preferred term coded according to the MedDRA dictionary. Tabulations will be by subject, such that subjects are only counted once within each body system or preferred term. These summaries will be provided for the following:

- all TEAEs, and the total number of events reported
- TEAEs of special interest
- TEAEs related to study treatment (i.e. Related or Possibly Related)
- TEAEs with Grade ≥3 (severe)
- TEAEs leading to study discontinuation
- Serious TEAE's
- TEAEs resulting in death

All adverse events (including non-treatment-emergent events) recorded on the CRF will be listed.

Rash assessments will be listed separately for subjects with this AESI.


#### 12.8.2 Deaths and Serious Adverse Events

A listing of all deaths that occurred following the first dose of treatment will be presented in a listing. Similarly, all AEs noted as serious will be displayed in a listing.

#### 12.8.3 Central Laboratory Data

Laboratory data will be summarized in the Safety Population using descriptive statistics (based on SI units) for the observed and change from baseline results for hematology and clinical chemistry by treatment group at each visit. Only the numeric part in laboratory values that contain non-numeric qualifiers, such as less than (<) a certain value, or greater than (>) a certain value, will be used in the summary statistics.

For continuous data, the following hematology tests will be summarized for observed and change from baseline values:

 Basophils (% and abs), Blasts (% and abs), Eosinophils (% and abs), Hematocrit, Hemoglobin, Lymphocytes (% and abs), mean corpuscular hemoglobin concentration (MCHC), mean corpuscular volume (MCV), Monocytes (% and abs), Neutrophils (% and abs), Platelets, red blood cell (RBC) count, RBC Morphology, Reticulocyte Count (% and abs), white blood cell (WBC) count

The following chemistry tests will be summarized for observed and change from baseline values:

 Alkaline Phosphatase, Albumin, ALT (SGPT), Amylase, AST (SGOT), Bicarbonate, Bilirubin (direct), Bilirubin (indirect), Bilirubin (total), Calcium, Chloride, Cholesterol, Creatinine, estimated GFR (eGFR) CKD, GGT, Globulin, lactate dehydrogenase (LDH), Lipase, Phosphorus, Potassium, Serum Glucose, Sodium, Total Protein, Triglycerides, Urea Nitrogen (BUN), Uric Acid

The following coagulation factors will be summarized for observed and change from baseline values:

 International normalized ratio (INR), Prothrombin time (PT) and activated partial thromboplastin time (aPTT).

The following urinalysis parameters will be summarized for observed and change from baseline values:

- Continuous parameters: pH, Specific gravity
- Categorical parameters: protein, glucose, ketones, blood

Clinically abnormal laboratory values will be applied based on the modified Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences (2017), as noted in <u>Appendix 3</u>. In the summary tables, values of grading will be displayed as 0, 1, 2, 3, or 4, where a grade of '0' will be assigned if the lab value was non-missing but did not meet a grading criterion (i.e. defined as normal). The maximum post-baseline grade observed up to end of study will be tabulated for each laboratory test, and percentages will be based on the number of subjects with a post-baseline evaluation of the specific laboratory test.

Additionally, a shift table will be used to tabulate the grading observed at Baseline to the maximum post-Baseline result up to the end of study for each lab parameter, in order to highlight important grading differences noted during the study.

The DAIDS grades will be applied within the Covance central lab datasets for the following parameters:

Hematology: Hemoglobin, Lymphocytes (absolute), Neutrophils (absolute), Platelets, and WBC.


 Chemistry: Alkaline Phosphatase, Albumin, ALT (SGPT), Amylase, AST (SGOT), Bicarbonate, Bilirubin (total), Calcium, Creatinine, eGFR CKD, GGT, Lipase, Phosphorus, Potassium, Serum Glucose, Sodium, Uric Acid

· Coagulation: PT, aPTT, and INR

For subjects reporting an AESI of ALT Flare, a separate summary lab data associated with the flare will be presented for both treatment groups. Data may include results for clinical chemistries (i.e. AST, ALT, GGT, alkaline phosphatase, total bilirubin, and albumin).

For subjects with abnormal ALT at Baseline (defined as modified DAIDS grading of ≥ 1), the number and percentage of subjects who have normal ALT at Week 24 (i.e. a grading of 0) will be presented.

A shift table will be used to tabulate the ALT levels observed at baseline to post-baseline measurements up to end of the study for the following categories: Normal (ALT < ULN), ALT >= 1xULN to < 3xULN, ALT >= 3xULN to < 5xULN, ALT >= 5xULN to < 20xULN, ALT >= 20xULN.By-patient listings will be provided for hematology, clinical chemistry, coagulation, and urinalysis. Laboratory values outside normal limits will be identified in the subject data listings with flags for low (L) and high (H).

Additional listings will be provided for other laboratory assessments, including serum alpha fetoprotein (AFP), hemoglobin A1c (HbA1c), and follicle-stimulating hormone (FSH; females only) as collected, as well as information collected regarding drug abuse from the urine drug results (i.e. amphetamine, barbiturates, benzodiazepines, cannabinoids, cocaine, propoxyphene, ethanol, opiates, and phencyclidine).

Antibody tests for hepatitis B surface antigen (HBsAb), hepatitis B "e" antigen (HBeAb), hepatitis C virus (HCV), hepatitis D virus (HDV), hepatitis A virus immunoglobulin M (HAV IgM), hepatitis E virus immunoglobulin M (HEV IgM), HBV core protein (HBCrAb), and human immunodeficiency virus (HIV) will be listed by subject as collected.

#### 12.8.4 Vital Signs

Blood pressure (systolic and diastolic), respiratory rate (breaths/min), pulse rate (beats/min), and temperature (°C) will be summarized in the Safety Population using descriptive statistics, for both the absolute and the change from baseline assessments over time. Timepoints will include screening, Baseline (Day 1), and Weeks 2, 4, 8, 12, 16, 20, and 24, and follow-up samples will be collected Weeks 28 and 36 for subjects who do not continue treatment in the extension protocol. Weight (kg) will also be included in the summary table, for the following timepoints: Screening, Baseline (Day 1), and Weeks 4, 24, and Week 36 for subjects who remain in the follow-up period.

#### 12.8.5 Physical Examinations, ECGs, and Other Observations Related to Safety

Physical examination results will be summarized in the Safety Population by body system for each timepoint based on the frequency and percentage of subjects with interpretations of normal, abnormal – clinically significant, abnormal – not clinically significant, or not done. Results of 12-lead ECG interpretations will be presented by timepoint in a similar manner.

For female subjects in the Safety Population, results from blood (serum  $\beta$ -hCG) and urine pregnancy tests will be tabulated. All results will be presented in a data listing.

#### 12.9 Pharmacokinetics

For ABI-H0731-treated subjects with a PK assessment (i.e. subjects in Pharmacokinetic Set 1), summary statistics will be presented for trough PK plasma concentrations observed at Baseline, Weeks 2, 4, 12, and

PRS 005 T 17 G 

Statistical Analysis Plan


24, as well as Week 28 for subjects who enter the follow-up phase. If a subject consents to optional post-dose PK sample collections, then the post-dose (peak) concentration, and the trough to peak ratio will be summarized descriptively at Baseline, Week 2 and Week 4.

For all subjects receiving ETV with a PK assessment (i.e. subjects in Pharmacokinetic Set 2), a similar analysis as described above will be provided, for both treatment groups.

For subjects in Pharmacokinetic Set 2 (treated with ETV), the comparison of ETV trough concentration between treatment arms (ABI-H0731 vs Placebo) will be presented in a table. The comparison will be based on the geometric mean ratio (with 90% CI) obtained from a two-sample t-test that compares the natural log-transformed trough PK measurements between treatment arms.

Trough plasma concentrations for ETV levels in subjects randomized to ABI-H0731 vs Placebo at Baseline, Week 2, Week 4, Week 12, and Week 24, as well as Week 28 (for subjects who enter the follow-up phase) will be presented side-by-side in a graph. At each timepoint, the following results will be plotted: ETV PK levels in ABI-H0731 subjects, and ETV PK levels in Placebo subjects.

Drug-drug interaction effects of ETV at Baseline, Week 2, Week 4, Week 12, Week 24, and Week 28 (for subjects who enter the follow-up phase) will be presented in a graph. At each time point the geometric mean ratio of trough ETV PK values for [ABI-H0731 + ETV / ETV alone] will be plotted.

#### 13.0 Validation

PRA's goal is to ensure that each TFL delivery is submitted to the highest level of quality. Our quality control procedures will be documented separately.

#### 14.0 References

None.



Statistical Analysis Plan


## **Appendix 1 Glossary of Abbreviations**

| Classary of Abbreviations | |
|---|---|
| Glossary of Abbreviations | |
| AE | adverse event |
| AESI | adverse event of special interest |
| AFP | alpha fetoprotein |
| ALT | alanine aminotransferase |
| aPTT | activated partial thromboplastin time |
| AST | aspartate aminotransferase |
| ATC | Anatomic therapeutic classification |
| AUC | area under the concentration-time curve |
| BMI | body mass index |
| cccDNA | covalently closed circular DNA |
| CHB | chronic hepatitis B infection |
| CKD-EPI | Chronic Kidney Disease Epidemiology Collaboration |
| CI | confidence interval |
| CRF | case report form |
| CRO | Clinical Research Organization (PRA Health Sciences) |
| CTMS | Clinical Trials Management System (PRA) |
| DAIDS | Division of AIDS |
| DMC | Data Monitoring Committee |
| dsDNA | double-stranded DNA |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| eGFR | estimated glomerular filtration rate |
| ETV | entecavir |
| FSH | follicle-stimulating hormone |
| GFR | glomerular filtration rate |
| HAV | hepatitis A virus |
| HbA1c | hemoglobin A1c |
| HBCrAb | antibody to the HBV core protein |
| HBCrAg | hepatitis B core-related antigen |
| HBeAb | HBeAg antibody |
| HBeAg | hepatitis B "e" antigen |
| HBsAb | HBsAg antibody |
| HBsAg | hepatitis B surface antigen |
| HBV | hepatitis B virus |
| HCV | hepatitis C virus |
| HDV | hepatitis D virus |
| HEV | hepatitis E virus |
| HIV | ' |
| ICF | human immunodeficiency virus Informed Consent Form |
| IgM | immunoglobulin M |
| INR | International Normalized Ratio |
| ITT | Internetive Web Response System |
| IWRS | Interactive Web Response System |
| LOQ | limit of quantitation |
| MCHC | mean corpuscular hemoglobin concentration |

PRS 005 T 17 G 



Statistical Analysis Plan


| II. | <u>`</u> |
|---|---|
| MCV | mean corpuscular volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | magnetic resonance imaging |
| NUC | nucleos(t)ide inhibitors of the HBV polymerase; also called nucleos(t)ide analogues or nucleos(t)ides |
| PG | pharmacogenomic |
| pgRNA | pre-genomic RNA |
| PK | pharmacokinetic(s) |
| PK1 | Pharmacokinetic Population 1 |
| PK2 | Pharmacokinetic Population 2 |
| PT | prothrombin time |
| rcDNA | relaxed circular DNA |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SOC | standard of care |
| TAF | tenofovir alafenamide |
| TDF | tenofovir disoproxil fumarate |
| TEAE | treatment-emergent adverse event |
| TFL | tables, figures, and listings |
| ULN | upper limit of normal |
| WHO | World Health Organization |

Statistical Analysis Plan


# Appendix 2 Tables, Figures, Listings, and Supportive SAS Output Appendices

Please refer to the Table, Figure and Listing shells to support this SAP, provided in a separate document.

Isolated missing values will be imputed by Markov Chain Monte Carlo (SAS PROC MI, MCMC) first to make the missing pattern monotone and then imputed by monotone linear regression. SAS PROC MI and PROC MIXED will be used to obtain MMRM estimates of treatment difference. SAS PROC MIANALYZE will be used to combine estimates and to generate the average test statistics for hypothesis testing. The Missing at Random method will be used with the following parameters: MAR — assume missing at random, number of imputation=100, seed= SEED11 (for MCMC) and SEED12 (for MONOTONE REG) for imputation.

PRS 005 T 17 G 


## **Appendix 3 Grading of Laboratory Values**

TOXICITY GRADING OF LABORATORY ABNORMALITIES AND CLINICAL ADVERSE EVENTS. PUBLISH DATE: JULY 2017

Adapted from the U.S. National Institutes of Health (Division of AIDS) Table for Grading Severity of Adult Adverse Experiences (2017). Parameters within the table that have been modified for this study are designated by an asterisk (\*).



Statistical Analysis Plan


## **Laboratory Values\*: Chemistries**

| Laboratory Valu | Laboratory Values*: Chemistries | | | |
|---|---|---|---|---|
| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
| Acidosis | NA | pH≤7.3 to <lln< td=""><td>pH&lt;7.3 without life-<br/>threatening<br/>consequences</td><td>pH&lt;7.3 with life-<br/>threatening<br/>consequences</td></lln<> | pH<7.3 without life-<br>threatening<br>consequences | pH<7.3 with life-<br>threatening<br>consequences |
| Albumin, Low | 3.0 to < LLN | $\geq$ 2.0 to $<$ 3.0 | < 2.0 | NA |
| (g/dL; g/L) | 30 to < LLN | $\geq$ 20 to < 30 | < 20 | |
| Alkaline<br>Phosphatase, High | 1.25 to < 2.5 x ULN | 2.5 to < 5.0 x ULN | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Alkalosis | NA | pH > ULN to $\leq 7.5$ | pH > 7.5 without life-<br>threatening<br>consequences | pH > 7.5 with life-<br>threatening<br>consequences |
| ALT or SGPT, High Report only one | 1.25 to < 2.5 x ULN | 2.5 to < 5.0 x ULN | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Amylase<br>(Pancreatic) or<br>Amylase (Total),<br>High Report only one | 1.1 to <1.5×ULN | 1.5 to <3.0×ULN | 3.0 to <5.0×ULN | ≥5.0×ULN |
| AST or SGOT, High Report only one | 1.25 to < 2.5 x ULN | 2.5 to < 5.0 x ULN | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Bicarbonate, Low (mEq/L; mmol/L) | 16.0 to <lln 16.0="" <lln<="" td="" to=""><td>11.0 to &lt;16.0 <i>11.0 to</i> &lt;16.0</td><td>8.0 to &lt;11.0<br/>8.0 to &lt;11.0</td><td>&lt;8.0<br/>&lt;8.0</td></lln> | 11.0 to <16.0 <i>11.0 to</i> <16.0 | 8.0 to <11.0<br>8.0 to <11.0 | <8.0<br><8.0 |
| Bilirubin<br>Direct Bilirubinm,<br>High | NA | NA | >ULN with other signs and symptoms of hepatotoxicity. | >ULN with life-<br>threatening<br>consequences (e.g.,<br>signs and symptoms of<br>liver failure) |
| Total Bilirubin, High | 1.1 to <1.6×ULN | 1.6 to <2.6×ULN | 2.6 to <5.0×ULN | ≥5.0×ULN |
| Calcium, High (mg/dL; mmol/L) | 10.6 to <11.5<br>2.65 to <2.88 | 11.5 to <12.5<br>2.88 to <3.13 | 12.5 to <13.5<br>3.13 to <3.38 | ≥13.5<br>≥3.38 |
| Calcium (Ionized),<br>High (mg/dL;<br>mmol/L) | >ULN to <6.0<br>>ULN to <1.5 | 6.0 to <6.4<br>1.5 to <1.6 | 6.4 to <7.2<br>1.6 to <1.8 | ≥7.2<br>≥1.8 |
| Calcium, Low (mg/dL; mmol/L) | 7.8 to <8.4<br>1.95 to <2.10 | 7.0 to <7.8<br>1.75 to <1.95 | 6.1 to <7.0<br>1.53 to <1.75 | <6.1<br><1.53 |
| Calcium (Ionized),<br>Low (mg/dL;<br>mmol/L) | <lln 4.0<br="" to=""><lln 1.0<="" td="" to=""><td>3.6 to &lt;4.0<br/>0.9 to &lt;1.0</td><td>3.2 to &lt;3.6<br/>0.8 to &lt;0.9</td><td>&lt;3.2<br/>&lt;0.8</td></lln></lln> | 3.6 to <4.0<br>0.9 to <1.0 | 3.2 to <3.6<br>0.8 to <0.9 | <3.2<br><0.8 |
| Cardiac Troponin I,<br>High | NA | NA | NA | Levels consistent with<br>myocardial infarction<br>or unstable angina as<br>defined by the local<br>laboratory |
| Creatine Kinase,<br>High | 3 to <6×ULN | 6 to <10×ULN | 10 to <20×ULN | ≥20×ULN |
| Creatinine, High<br>*Report only one | 1.1 to 1.3×ULN | >1.3 to 1.8×ULN OR<br>Increase to 1.3 to<br><1.5×participant's<br>baseline | >1.8 to <3.5×ULN OR<br>Increase to 1.5 to<br><2.0×participant's<br>baseline | ≥3.5×ULN OR Increase of ≥2.0×participant's baseline |

PRS 005 T 17 G 

Statistical Analysis Plan


#### **Laboratory Values\*: Chemistries**

| · | Carlo 1 Mil | | G 1- 2 G | Grade 4 Potentially |
|---|---|---|---|---|
| Parameter Creatinine Clearance 13 or eGFR, Low *Report only one | NA NA | Grade 2 Moderate <90 to 60 ml/min or ml/min/1.73 m² OR 10 to <30% decrease from participant's baseline | Grade 3 Severe <60 to 30 ml/min or ml/min/1.73 m² OR 30 to <50% decrease from participant's baseline | <pre>&lt;30 ml/min or ml/min/1.73 m² OR ≥50% decrease from participant's baseline</pre> |
| Glucose (mg/dL;<br>mmol/L) Fasting,<br>High | 110 to 125<br>6.11 to <6.95 | >125 to 250<br>6.95 to <13.89 | >250 to 500<br>13.89 to <27.75 | or dialysis needed<br>≥500<br>≥27.75 |
| Nonfasting, High | 116 to 160 | >160 to 250 | >250 to 500 | ≥500 |
| | 6.44 to <8.89 | 8.89 to <13.89 | 13.89 to <27.75 | ≥27.75 |
| Glucose, Low (mg/dL; mmol/L) | 55 to 64 | 40 to <55 | 30 to <40 | <30 |
| | 3.05 to <3.55 | 2.22 to <3.05 | 1.67 to <2.22 | <1.67 |
| Lactate, High | ULN to <2.0×ULN without acidosis | ≥2.0×ULN without acidosis | Increased lactate with pH <7.3 without life-threatening consequences | Increased lactate with pH <7.3 with life-threatening consequences |
| Lipase, High | 1.1 to <1.5×ULN | 1.5 to <3.0×ULN | 3.0 to <5.0×ULN | ≥5.0×ULN |
| Lipid Disorders (mg/dL; mmol/L) | 200 to <240 | 240 to <300 | ≥300 | NA |
| Cholesterol, Fasting,<br>High | 5.18 to <6.19 | 6.19 to <7.77 | ≥7.77 | |
| LDL, Fasting, High | 130 to <160<br>3.37 to <4.12 | 160 to <190<br>4.12 to <4.90 | ≥190<br>≥4.90 | NA |
| Triglycerides, | 150 to 300 | >300 to 500 | >500 to <1,000 | >1,000 |
| Fasting, High | 1.71 to 3.42 | >3.42 to 5.7 | >5.7 to 11.4 | >11.4 |
| Magnesium <sup>14</sup> , Low (mEq/L; mmol/L) | 1.2 to <1.4 | 0.9 to <1.2 | 0.6 to <0.9 | <0.6 |
| | 0.60 to <0.70 | 0.45 to <0.60 | 0.30 to <0.45 | <0.30 |
| Phosphate (Phosphorus), Low (mg/dL; mmol/L) | 2.0 to <lln< td=""><td>1.4 to &lt;2.0</td><td>1.0 to &lt;1.4</td><td>&lt;1.0</td></lln<> | 1.4 to <2.0 | 1.0 to <1.4 | <1.0 |
| | 0.65 to <lln< td=""><td>0.45 to &lt;0.65</td><td>0.32 to &lt;0.45</td><td>&lt;0.32</td></lln<> | 0.45 to <0.65 | 0.32 to <0.45 | <0.32 |
| Potassium, High (mEq/L; mmol/L) | 5.6 to <6.0 | 6.0 to <6.5 | 6.5 to <7.0 | ≥7.0 |
| | 5.6 to <6.0 | 6.0 to <6.5 | 6.5 to <7.0 | ≥7.0 |
| Potassium, Low (mEq/L; mmol/L) | 3.0 to <3.4 | 2.5 to <3.0 | 2.0 to <2.5 | <2.0 |
| | 3.0 to <3.4 | 2.5 to <3.0 | 2.0 to <2.5 | <2.0 |
| Sodium, High | 146 to <150 | 150 to <154 | 154 to <160 | ≥160 |
| (mEq/L; mmol/L) | 146 to <150 | 150 to <154 | 154 to <160 | ≥160 |
| Sodium, Low (mEq/L; mmol/L) | 130 to <135 | 125 to <130 | 121 to <125 | ≤120 |
| | 130 to <135 | 125 to <130 | 121 to <125 | ≤120 |
| Uric Acid, High (mg/dL; mmol/L) | 7.5 to <10.0 | 10.0 to <12.0 | 12.0 to <15.0 | ≥15.0 |
| | 0.45 to <0.59 | 0.59 to <0.71 | 0.71 to <0.89 | ≥0.89 |

<sup>\*</sup>Reminder: Choose the method that selects for the higher grade.

<sup>\*</sup>Reminder: An asymptomatic abnormal laboratory finding without an accompanying adverse event should not be reported to DAIDS in an expedited time frame unless it meets protocol-specific reporting requirements.

<sup>13</sup> Use the applicable formula (i.e., Cockcroft-Gault in mL/min or Schwartz, MDRD, CKD-Epi in mL/min/1.73m²). Sites should choose the method defined in their study and when not specified, use the method most relevant to the study population.

<sup>14</sup> To convert a magnesium value from mg/dL to mmol/L, laboratories should multiply by 0.4114.

Statistical Analysis Plan


#### Hematology

| Hematology | I | 1 | 1 | |
|---|---|---|---|---|
| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
| Absolute CD4+ Count, Low (cell/mm³; cells/L) (not HIV infected) | 300 to <400<br>300 to <400 | 200 to <300<br>200 to <300 | 100 to <200<br>100 to <200 | <100<br><100 |
| Absolute Lymphocyte<br>Count, Low<br>(cell/mm³; cells/L)<br>(not HIV infected) | 600 to <650<br>0.600×10 <sup>9</sup> to<br><0.650×10 <sup>9</sup> | 500 to <600<br>0.500×10 <sup>9</sup> to<br><0.600×10 <sup>9</sup> | 350 to <500<br>0.350×10 <sup>9</sup> to<br><0.500×10 <sup>9</sup> | <350<br><0.350×10 <sup>9</sup> |
| Absolute Neutrophil<br>Count (ANC), Low<br>(cells/mm³; cells/L) | 800 to 1,000<br>0.800×10 <sup>9</sup> to<br>1.000×10 <sup>9</sup> | 600 to 799<br>0.600×10 <sup>9</sup> to<br>0.799×10 <sup>9</sup> | 400 to 599<br>0.400×10 <sup>9</sup> to<br>0.599×10 <sup>9</sup> | <400<br><0.400×10 <sup>9</sup> |
| Fibrinogen, Decreased (mg/dL; g/L) | 100 to <200<br>1.00 to <2.00 OR 0.75<br>to <1.00×LLN | 75 to <100<br>0.75 to <1.00 OR<br>≥0.50 to <0.75×LLN | 50 to <75<br>0.50 to <0.75 OR<br>0.25 to <0.50×LLN | <50<br><0.50 OR<br><0.25×LLN OR<br>Associated with gross<br>bleeding |
| Hemoglobin <sup>15</sup> , Low<br>(g/dL; mmol/L) <sup>16</sup><br>Male only | 10.0 to 10.9<br>6.19 to 6.76 | 9.0 to <10.0<br>5.57 to <6.19 | 7.0 to <9.0<br>4.34 to <5.57 | <7.0<br><4.34 |
| Hemoglobin <sup>15</sup> , Low (g/dL; mmol/L) <sup>16</sup> female only | 9.5 to 10.4<br>5.88 to 6.48 | 8.5 to <9.5<br>5.25 to <5.88 | 6.5 to <8.5<br>4.03 to <5.25 | <6.5<br><4.03 |
| INR, High (not on<br>anticoagulation<br>therapy) | 1.1 to <1.5×ULN | 1.5 to <2.0×ULN | 2.0 to <3.0×ULN | ≥3.0×ULN |
| Methemoglobin (% hemoglobin) | 5.0 to <10.0% | 10.0 to <15.0% | 15.0 to <20.0% | ≥20.0% |
| PTT, High (not on anticoagulation therapy) | 1.1 to <1.66×ULN | 1.66 to <2.33×ULN | 2.33 to <3.00×ULN | ≥3.00×ULN |
| Platelets, Decreased (cells/mm³; cells/L) | 100,000 to <125,000<br>100.000×10 <sup>9</sup> to<br><125.000×10 <sup>9</sup> | 50,000 to <100,000<br>50.000×10 <sup>9</sup> to<br><100.000×10 <sup>9</sup> | 25,000 to <50,000<br>25.000×10 <sup>9</sup> to<br><50.000×10 <sup>9</sup> | <25,000<br><25.000×10 <sup>9</sup> |
| PT, High<br>(not on anticoagulation<br>therapy) | 1.1 to <1.25×ULN | 1.25 to <1.50×ULN | 1.50 to <3.00×ULN | ≥3.00×ULN |
| WBC, Decreased (cells/mm³; cells/L) | 2,000 to 2,499<br>2.000×10 <sup>9</sup> to<br>2.499×10 <sup>9</sup> | 1,500 to 1,999<br>1.500×10 <sup>9</sup> to<br>1.999×10 <sup>9</sup> | 1,000 to 1,499<br>1.000×10 <sup>9</sup> to<br>1.499×10 <sup>9</sup> | <1,000<br><1.000×10 <sup>9</sup> |

<sup>15</sup> Male and female sex are defined as sex at birth. For transgender participants who have been on hormone therapy for more than 6 consecutive months, grade hemoglobin based on the gender with which they identify (i.e., a transgender female should be graded using the female sex at birth hemoglobin laboratory values).

PRS 005 T 17 G 

<sup>16</sup> The most commonly used conversion factor to convert g/dL to mmol/L is 0.6206. For grading hemoglobin results obtained by an analytic method with a conversion factor other than 0.6206, the result must be converted to g/dL using appropriate conversion factor for the particular laboratory.



Statistical Analysis Plan


## Urinalysis

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Glycosuria (random collection tested by dipstick) | Trace to 1+ or ≤250 mg | 2+ or >250 to ≤500 mg | >2+ or >500 mg | NA |
| Hematuria (not to be<br>reported based on<br>dipstick findings or on<br>blood believed to be<br>of menstrual origin) | 6 to <10 RBCs per<br>high power field | ≥10 RBCs per high<br>power field | Gross, with or without<br>clots OR With RBC<br>casts OR Intervention<br>indicated | Life-threatening consequences |
| Proteinuria (random collection tested by dipstick) | 1+ | 2+ | 3+ or higher | NA |